CLINICAL TRIAL: NCT07065097
Title: Impact an Educational Multimodal Intervention to Improve Healthy Habits in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Dr. Fidel Lopez Espuela, PhD Psicologist, Nurse Registered, University of Extremadura
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UExtremadura2020
Record Dates: First submitted 2024-08-29; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2024-08

CONDITIONS: Diet, Healthy; Adolescent Overweight; Child Nutrition Sciences; Exercise; Self Concept; Body Dissatisfaction
Keywords: Diet, Healthy; Adolescent; Physical Activity; Exercise; self concept; body image
MeSH Terms: conditions — Pediatric Obesity; Motor Activity | interventions — Nutritional Status

STUDY DESIGN:
Intervention Model Description: Controlled and intervention
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No intervention
- Intervention group (Experimental): This group underwent a multimodal intervention in which they worked on self-esteem, self-concept and body image.
  Interventions: Other: A multimodal intervention in which they worked on self-esteem, self-concept and body image and nutrition.

INTERVENTIONS:
Other: A multimodal intervention in which they worked on self-esteem, self-concept and body image and nutrition. — A multimodal intervention in which they worked on self-esteem, self-concept and body image and nutrition.
  Arms: Intervention group

SUMMARY:
Background:

Adolescence is a critical period to promote healthy habits.

Objective: To know the impact that a multimodal educational intervention has on the knowledge and modification of healthy habits (HS) (Mediterranean diet (DM) and physical activity) in adolescents.

Methodology: randomized controlled clinical trial, with multimodal educational intervention, in the Diocesan College of Cáceres.

The participants will be assign to the control (GC) or experimental (GE) group by randomization, the latter received a multimodal educational intervention (theoretical and practical workshops on HS).

Data will be collect: sociodemographic, academic notes, anthropometric data, KIDMED questionnaire and physical activity questionnaire (PAQ-A); Pre and post intervention. And knowledge about HS will be evaluate.

The parents of the intervention group will receive workshops on healthy habits, benefits of diet and physical exercise, as well as the adolescents of the intervention group.

All parents will grant consent to participate.

ELIGIBILITY:
. Inclusion Criteria:

• aged between 11 and 16 years who were in their 1st and 2nd years of compulsory secondary education (ESO).

Exclusion Criteria:

* adolescents with serious illnesses such as cancer or with serious mental health problems (depression requiring treatment) and
* Adolescents who, despite having parental consent, did not wish to participate.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 385 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Self steem | 4 months
  Self-esteem was assessed with the Rosenberg Scale. consists of 10 items and is a self-report instrument for evaluating an individual's overall self-esteem. The RSES is scored using four response options, ranging from strongly agree to strongly disagree. It is a two-dimensional scale: positive self-esteem (self-confidence or personal satisfaction) and negative self-esteem (self-contempt or personal devaluation). Five items are scored positively, and five items are scored negatively. The total score ranges from 10 to 40 points, with 10 points being the lowest self-esteem score and 40 points being the highest. With respect to the total score, a score of 30 to 40 points indicates high self-esteem; a score of 26 to 29 points indicates intermediate self-esteem; and a score less than or equal to 25 points indicate low self-esteem.
Body image | 4 months
  Dissatisfaction with body image was assessed with the Body shape questionnaire. This instrument evaluates dissatisfaction with body image due to body weight and shape; participants respond to items referring to how they have felt about their body shape in the last weeks. The questionnaire contains 34 self-report items; items are scored using a six-point Likert scale ranging from 1 (never) to 6 (always), with a total possible score ranging from 34 to 204 points. The higher the score is, the greater an individual's dissatisfaction with their body. Based on their BSQ results, the participants were divided into four groups according to dissatisfaction with physical appearance using the validated model: scores ≤80 (no dissatisfaction with BI); 81 ≤ scores ≤ 110 (slight dissatisfaction with BI); 111≤ scores ≤ 140 (moderate dissatisfaction with BI); and scores ≥ 141 (severe dissatisfaction with BI).
self concept | 4 months
  self-concept was assessed with the physical self-concept questionnaire.
  The Physical Activity Questionnaire for Adolescents (PAQ-A) assesses the physical exercise of the adolescent in the last 7 days. It consists of 9 questions that measure aspects of the physical exercise performed by the adolescent. It also provides information on whether the person has been ill. It is evaluated by means of a scale of 1 to 5 points that establishes a graduation of the level of physical activity carried out. It allows us to know at what time of the day and of the week the adolescent is most active.
Nutrition | 4 months
  the quality of the diet was assessed with the kidmed questionnaire. Kidmed questionnaire assesses adherence to the Mediterranean diet as a prototype of a healthy diet. The index consists of 16 questions, of which 12 are positive and 4 are negative; individuals who answer "yes" to positive questions receive +1 point, while those who answer "yes" to negative questions receive -1 point. Points are summed at the end of the evaluation, and a score ranging from 0 to 12 is obtained. The sum of these value scores is classified into 3 levels: ≥8 points indicates the optimal Mediterranean diet (good), scores between 4 and 7 points indicate that compatibility with the Mediterranean diet should be improved (moderate), and scores ≤3 points indicate very poor diet quality (low)

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Nursing and Ocupational Therapy College. University of Extremadura, Cáceres, Caceres
  - Nursing and Ocupational Therapy College. University of Extremadura, Cáceres, CÁCERES

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benitez-Sillero JD, Portela-Pino I, Morente A, Raya-Gonzalez J. Longitudinal Relationships Between Physical Fitness With Physical Self-Concept and Self-Esteem in Adolescents. Res Q Exerc Sport. 2024 Mar;95(1):183-189. doi: 10.1080/02701367.2023.2173134. Epub 2023 Apr 10. PMID 37036415